CLINICAL TRIAL: NCT00776945
Title: Determine the Feasibility and Functionality of fPAM Imaging for the in Vivo Characterization and Early Diagnosis of Melanoma
Brief Title: Feasibility and Functionality of fPAM Imaging in Melanoma
Acronym: fPAM
Status: Terminated | Type: Observational
Why Stopped: no funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Lynn Cornelius, MD, Chief, Division of Dermatology, Washington University School of Medicine
Other Study IDs: 07-0635
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2013-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue biopsies may be performed if locoregional recurrence validated by clinical examination.
Oversight: Data Monitoring Committee: No

SUMMARY:
Melanoma is a cutaneous malignancy that has the potential for local (skin) and regional (lymph node) recurrence. These recurrences may be difficult to detect in their earliest stages. We are attempting to use novel form of skin imaging that uses ultrasound combined with laser to identify these recurrences early, when they may be most amenable to treatment. This imaging will detect melanoma pigment below the surface of the skin and in the draining lymph nodes, as well as new blood vessel formation that occurs with these loco-regional metastases.

DETAILED DESCRIPTION:
recruiting healthy individuals with pigmented lesions and individuals with melanoma and pigmented lesions

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 yrs of age) with recently diagnosed or a history of, Stage I - III melanoma who are able to give informed consent.

Exclusion Criteria:

* Patients with melanomas < 1mm.
* Pregnant females.
* Children and young adults < 18 yrs of age and patients who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage I - III melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
fPAM is a hybrid imaging technique that detects absorbed diffuse photons ultrasonically through the photoacoustic (PA) effect | baseline
  Evaluate pigmented lesions for depth, width, total hemoglobin saturation, melanin distribution, and melanin concentration using fPAM in vivo and ex vivo

CONTACTS AND LOCATIONS:
Overall Officials: Lynn A Cornelius, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri